CLINICAL TRIAL: NCT00002195
Title: A Phase III Trial to Evaluate the Safety and Antiviral Efficacy of 141W94 in Combination With Retrovir and Epivir Compared to Retrovir and Epivir Alone in Patients With HIV Infection.
Brief Title: A Study of Retrovir and Epivir Alone or in Combination With 141W94 in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 264D; PROA3001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — amprenavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Amprenavir
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to see if it is safe and effective to add 141W94 to an anti-HIV regimen that includes retrovir plus epivir.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, two-arm study comparing treatment with a triple regimen consisting of 141W94, retrovir, and epivir and a double regimen consisting of retrovir and epivir.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-positive status.
* Screening viral load >= 10,000 copies/mm3 14 days prior to entry.
* CD4+ cell counts >= 200 cells/mm3 14 days prior to entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

Clinical diagnosis of AIDS (CDC 1993 Classification C).

Concurrent Medication:

Excluded:

Terfenadine, astemizole, cisapride, triazolam, medazolam, and ergotamine/dihydroergotamine-containing regimens.

Patients with the following prior conditions are excluded:

Clinically relevant hepatitis in the previous 6 months.

Prior Medication:

Excluded:

* Greater than 4 weeks of any nucleoside antiretroviral therapy.
* Previous therapy with an HIV protease inhibitor.
* Cytotoxic chemotherapeutic agents within 4 weeks prior to entry.
* Immunomodulating agents within 3 months prior to entry.

Prior Treatment:

Excluded:

Radiotherapy within 4 weeks prior to entry.

Risk Behavior:

Excluded:

Current alcohol or illicit drug use that may interfere with the patient's ability to comply with the dosing schedule or protocol evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Pacific Oaks Research, Beverly Hills, California
  - Dr Bruce Rashbaum, Washington D.C., District of Columbia
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - Community Research Initiative of Central Florida, Maitland, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Community Research Initiative of New England, Brookline, Massachusetts
  - Saint Vincent's AIDS Ctr, New York, New York
  - Methodist Hosp, Memphis, Tennessee